CLINICAL TRIAL: NCT05270798
Title: Triiodothyronine Hormone Supplementation Therapy in Patients With Septic Shock With Euthyroid Sick Syndrome
Brief Title: Thyroid Hormone Supplementation in Patients With Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cantonal Hospital Zenica (Other)
Responsible Party: Principal Investigator, Mirza Kovacevic, Anesthesiologist, Cantonal Hospital Zenica
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESS
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Euthyroid Sick Syndromes; Septic Shock
Keywords: septic shock; euthyroid sick syndrome; triiodothyronine
MeSH Terms: conditions — Euthyroid Sick Syndromes; Shock, Septic | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with low triiodothyronine levels who received triiodothyronine (Experimental)
  Interventions: Drug: triiodothyronine
- Patients with low triiodothyronine levels who received placebo (Placebo Comparator)
  Interventions: Drug: triiodothyronine
- Patients with low triiodothyronine and low tetraiodothyronine levels who received triiodothyronine (Experimental)
  Interventions: Drug: triiodothyronine
- Patients with low triiodothyronine and low tetraiodothyronine levels who received placebo (Placebo Comparator)
  Interventions: Drug: triiodothyronine

INTERVENTIONS:
Drug: triiodothyronine — Patients in septic shock who meet the diagnostic criteria for euthyroid sick syndrome will be divided into two groups; patients with low T3 levels and patients with low T3 and T4 levels. Both of these groups will be further randomly divided into patients receiving T3 hormone and patients receiving placebo.

SUMMARY:
The primary aim of the study would be to determine whether there is a difference in survival in the Intensive Care Unit between the group of patients with septic shock diagnosed with euthyroid sick syndrome who were treated with T3 hormone compared to the group of patients not treated with this hormone. Secondary objectives of the research would be:

Compare the level of thyroid hormones between the examined groups and

1. laboratory indicators of septic shock (C-reactive protein-CRP, procalcitonin, leukocytes, acid-base status, lactates)
2. APACHE II, SOFA and SAPS II patient assessment scales,
3. inflammatory prognostic systems (ratio of CRP and albumin-modified Glasgow prognostic score-mGPS, ratio of neutrophils and lymphocytes - NLR, ratio of platelets and lymphocytes - PLR, and ratio of leukocytes and CRP, prognostic index - PI)
4. hemodynamic stability of patients (MAP, systolic and diastolic pressure) in the periods of admission T0, T3, T6, T12, T24 and every 24 hours for 4 days,
5. effect of vasoactive drugs,
6. the need for mechanical ventilation categorized as yes or no, in case - number of respirator days,
7. length of stay in the Intensive Care Unit,
8. treatment outcome categorized as 28 day survival.

ELIGIBILITY:
Inclusion Criteria:

* all patients who meet the criteria for septic shock according to the definition of Surviving sepsis campaigning (The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA 2016): persistent hypotension requiring the use of vasoactive drugs to maintain mean arterial pressure ≥65 mm Hg ; blood lactates> 2 mmol / L despite adequate resuscitation volume,
* patients with laboratory-proven euthyroid sick syndrome, according to diagnostic criteria which include: normal levels of TSH hormone, low levels of T3 hormone that may accompany low levels of T4 hormone (depending on the stage of critical disease) and absence of previous primary thyroid and pituitary disease.

Exclusion Criteria:

* age below 18,
* patients with a history of thyroid disease or an enlarged thyroid gland,
* psychiatric patients,
* patients on hormone therapy (excluding insulin),
* those taking amiodarone, corticosteroids or dopamine
* pregnant or postpartum mothers 6 months ago,
* patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
The difference in survival in the Intensive Care Unit between the groups of patients with septic shock diagnosed with euthyroid sick syndrome who were treated with T3 hormone compared to the group of patients who were not treated with this hormone. | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital, Zenica, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kovacevic M, Adam VN, Causevic S. Triiodothyronine hormone supplementation therapy in septic shock patients with euthyroid sick syndrome: two pilot, placebo-controlled, randomized trials. Anaesth Crit Care Pain Med. 2024 Apr;43(2):101336. doi: 10.1016/j.accpm.2023.101336. Epub 2023 Dec 5. PMID 38061681